CLINICAL TRIAL: NCT03521037
Title: A Phase 1, Open-Label, Parallel Group Study to Determine the Pharmacokinetics, Safety and Tolerability of Rucaparib in Patients With an Advanced Solid Tumor and Either Moderate Hepatic Impairment or Normal Hepatic Function
Brief Title: Rucaparib Hepatic Impairment Study in Patients With a Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CO-338-078
Record Dates: First submitted 2018-02-14; First posted 2018-05-11 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Neoplasms
Keywords: rucaparib; CO-338; Clovis; Clovis Oncology; PARP inhibitor; hepatic impairment
MeSH Terms: conditions — Neoplasms | interventions — rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- no name (Experimental): Group 1: patients with normal hepatic function Group 2: patients who have moderate hepatic impairment
  Interventions: Drug: Rucaparib camsylate

INTERVENTIONS:
Drug: Rucaparib camsylate — In Part I, eligible patients will receive a single oral dose of 600 mg rucaparib followed by intensive plasma PK sampling up to Day 7 (hour 144). In Part II, patients may continue to receive continuous oral rucaparib in 28 day cycles.
  Other Names: rubraca

SUMMARY:
Phase 1, open-label, parallel group, PK, safety and tolerability study in patients with an advanced solid tumor and either normal hepatic function (Group 1, n = 8) or moderate hepatic impairment (Group 2, n = 8) according to the NCI-ODWG criteria. Patients in Group 1 and Group 2 may be enrolled in parallel, with preferential enrollment of Group 2 patients before Group 1 patients. The study will consist of 2 parts: a single-dose PK part (Part I) and a continuous rucaparib treatment part (Part II).

DETAILED DESCRIPTION:
In Part I, eligible patients will receive a single oral dose of 600 mg rucaparib followed by intensive plasma PK sampling up to Day 7 (hour 144). In Part II, patients may continue to receive continuous oral rucaparib in 28 day cycles. The starting dose for all Group 1 patients will be 600 mg BID. The first 2 patients with moderate hepatic impairment (Group 2) that enter Part II will receive a starting dose of 400 mg BID rucaparib; a lower dose of rucaparib may also be set based on PK results observed in Part I. If this initial starting dose is determined to be safe and tolerable as determined by real-time PK data and dose limiting toxicities (DLT) observed during the first 28 days of rucaparib, the starting dose of rucaparib may be increased in subsequent Group 2 patients. The starting dose for Group 2 patients may also be lowered, based on the patients' real time PK and emerging safety data. The Sponsor and key clinical research organization (CRO) staff will review available adverse event, laboratory, and PK data to determine the starting dose for subsequent Group 2 patients, as well as allowing intra-patient dose escalation of rucaparib after Cycle 1.Treatment with rucaparib will continue until progression of disease, unacceptable toxicity, death, loss to follow-up, withdrawal of consent, or other appropriate clinical reason for discontinuation.

ELIGIBILITY:
Inclusion Criteria:

All Patients:

* Patients ≥18 years of age at the time the ICF is signed;
* Patients with a histologically or cytologically confirmed advanced solid tumor who, in the opinion of the Investigator, could potentially benefit from treatment with rucaparib
* ECOG PS less than or equal to 2
* Adequate bone marrow and renal function

Hepatically Impaired Patients (in addition):

* Stable hepatic impairment as judged by the Investigator
* Moderate Hepatic Impairment (NCI-ODWG criteria) during Screening

Patients with Normal Hepatic Function (in addition):

• Normal Hepatic Function (NCI-ODWG criteria)

Exclusion Criteria:

All Patients:

* Prior treatment with chemotherapy, radiation, antibody therapy or other immunotherapy, gene therapy, vaccine therapy, angiogenesis inhibitors, or investigational drugs within 14 days prior to day 1
* Ongoing toxicity ≥ Grade 2 per Common Terminology Criteria for Adverse Events criteria (CTCAE version 4.03)
* Prior treatment with any poly adenosine diphosphate ribose polymerase inhibitor
* Arterial or venous thrombi (including cerebrovascular accident), myocardial infarction, admission for unstable angina, cardiac angioplasty, stenting or poorly controlled hypertension within the last 3 months prior to Screening
* Pre-existing duodenal stent, and/or any gastrointestinal disorder or defect that would, in the opinion of the Investigator, interfere with absorption of rucaparib
* Hospitalization for bowel obstruction within 3 months prior to Day 1
* Untreated or symptomatic central nervous system (CNS) metastases
* Evidence or history of bleeding disorder
* Acute illness within 14 days prior to Day 1
* Active second malignancy

Hepatically Impaired Patients (in addition):

* Severe hepatic encephalopathy (Grade >2);
* History of liver transplantation;
* Advanced ascites or ascites that require drainage and albumin supplementation, as judged by the Investigator;
* Acute damage of the liver with Grade 4 AST/ALT values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Maximum plasma rucaparib concentration (Cmax) | day 1 to day 7
  PK parameter of rucaparib to be calculated from the plasma concentration-time data
Area under the plasma rucaparib concentration-time curve from time zero up to the last time point with quantifiable concentration (AUC0-last) | day 1 to day 7
  PK parameter of rucaparib to be calculated from the plasma concentration-time data

SECONDARY OUTCOMES:
Area under the plasma rucaparib concentration-time curve from time zero up to time infinity (AUC0-inf) | day 1 to day 7
  PK parameter of rucaparib to be calculated from the plasma concentration-time data
Terminal half-life (t1/2) of rucaparib | day 1 to day 7
  PK parameter of rucaparib to be calculated from the plasma concentration-time data
Time to attain maximum plasma rucaparib concentration (Tmax) | day 1 to day 7
  PK parameter of rucaparib to be calculated from the plasma concentration-time data
Apparent clearance (CL/F) of rucaparib | day 1 to day 7
  PK parameter of rucaparib to be calculated from the plasma concentration-time data
Apparent volume of distribution during terminal phase (Vz/F) of rucaparib | day 1 to day 7
  PK parameter of rucaparib to be calculated from the plasma concentration-time data
Trough plasma concentration of rucaparib at steady state (Cmin,ss) | approximately 4 months
  PK parameter of rucaparib to be calculated from the plasma concentration-time data
Renal clearance (CLR) of rucaparib | day 1 to day 2
  PK parameter of rucaparib to be calculated from the plasma and urine concentration-time data
Cumulative amount of rucaparib excreted in urine during urine collection period post rucaparib dose | day 1 to day 2
  PK parameter of rucaparib to be calculated based on urine concentration-time data
Fraction of administered rucaparib excreted into urine (Fe/F) during urine collection period post rucaparib dose | day 1 to day 2
  PK parameter of rucaparib to be calculated based on the amount of rucaparib recovered in urine
Incidence of Adverse Events [Safety and Tolerability] | From Day 1 to last patient visit in Part II (approximately 2 years)
Incidence of clinical laboratory abnormalities [Safety and Tolerability] | From Day 1 to last patient visit in Part II (approximately 2 years)
Incidence of dose modifications [Safety and Tolerability] | From Day 1 to last patient visit in Part II (approximately 2 years)

OTHER OUTCOMES:
Maximum plasma metabolite concentration (Cmax) | day 1 to day 7
  PK parameter for rucaparib metabolite(s) to be calculated from plasma concentration-time data
Area under the plasma metabolite concentration-time curve from time zero up to the last time point with quantifiable concentrations (AUC0-last) | day 1 to day 7
  PK parameter for rucaparib metabolite(s) to be calculated from plasma concentration-time data
Area under the plasma metabolite concentration-time curve from time zero up to time infinity (AUC0-inf) | day 1 to day 7
  PK parameter for rucaparib metabolite(s) to be calculated from plasma concentration-time data
Terminal half-life (t1/2) of metabolite | day 1 to day 7
  PK parameter for rucaparib metabolite(s) to be calculated from plasma concentration-time data
Time to attain maximum plasma metabolite concentration (Tmax) | day 1 to day 7
  PK parameter for rucaparib metabolite(s) to be calculated from plasma concentration-time data
Plasma trough concentration of metabolite(s) at steady state (Cmin,ss) | day 1 to day 7
  PK parameter for rucaparib metabolite(s) to be calculated from plasma concentration-time data
Renal clearance (CLR) of metabolite(s) | day 1 to day 2
  PK parameters for rucaparib metabolite(s) to be calculated from plasma and urine concentration-time data
Cumulative amount of rucaparib metabolite(s) excreted in urine during urine collection period post rucaparib dose | day 1 to day 2
  PK parameter for rucaparib metabolite(s) to be calculated from urine concentration-time data

CONTACTS AND LOCATIONS:
Locations (6):
- Poland (4):
  - Wojewódzki Szpital Specjalistyczny w Białej Podlaskiej, Biała Podlaska
  - Med Polonia Sp. z o.o., Poznan
  - Zachodniopomorskie Centrum Onkologii w Szczecinie, Szczecin
  - BioVirtus Centrum Medyczne, Warsaw
- Summit Clinical Research s.r.o., Bratislava, Slovakia
- Northern Centre for Cancer Care, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No